CLINICAL TRIAL: NCT05112926
Title: Prospective, Single Arm Investigation to Assess Effectiveness and Safety of Embosphere Microspheres for Embolization of the Geniculate Artery for the Treatment of Pain With Known Moderate to Severe Knee Osteoarthritis
Brief Title: Effectiveness and Safety of Embosphere Microspheres for Embolization of the Geniculate Artery for the Treatment of Pain With Known Moderate to Severe Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Felipe Ferreira De Souza, Assistant Professor of Clinical Radiology, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20210848
Record Dates: First submitted 2021-11-01; First posted 2021-11-09 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Embosphere Microspheres group (Experimental): Participants in this group who are receiving standard of care (SOC) embolization surgery for the treatment of moderate to severe knee osteoarthritis will receive the Embospheres Microspheres during scheduled SOC surgery.
  Interventions: Device: Embosphere Microspheres

INTERVENTIONS:
Device: Embosphere Microspheres — Embosphere Microspheres are 100-300μm small, compressible, hydrophilic, biocompatible spheres made of acrylic polymer and porcine-derived gelatin used for embolization of geniculate artery.

SUMMARY:
The purpose of this research study is to evaluate the effectiveness and safety of a permanent embolic (Embosphere Microspheres) for embolization of the geniculate artery for the treatment of moderate to severe knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Subject has signed informed consent
* Subject is age 40-80
* Subject is able to have an MRI
* Minimum of prior 12 weeks of failed response to conservative therapy for knee osteoarthritis, which may include one or more of:

  a) Oral or topical NSAIDS, opioid medications, intra-articular injection of glucocorticoids or hyaluronic acid, physical therapy.
* Localized tenderness in anterior knee area
* Kellgren-Lawrence grade 1, 2, or 3 as assessed by weight-bearing knee radiographs
* Synovitis present as assessed by WORMS
* VAS >50 mm
* WOMAC score >30

Exclusion Criteria:

* Rheumatoid arthritis
* Local infection of the target knee(s)
* Kellgren-Lawrence grade >3
* Osteonecrosis evident by MRI
* Prior knee arthroplasty
* Allergy to iodinated contrast agents that cannot be managed by prophylaxis
* Hypersensitivity to gelatin products
* Any known condition that limits catheter-based intervention or is a contraindication to embolization
* Active malignancy other than non-melanomatous skin cancer
* Subject is pregnant, breastfeeding, or pre-menopausal and intending to become pregnant
* Any other condition related to the subject's health and wellbeing deemed exclusionary in the opinion of the investigator

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-12-08 (Actual); Primary Completion 2025-10-21 (Actual); Study Completion 2025-10-21 (Actual)

PRIMARY OUTCOMES:
Change in knee pain as assessed by the WOMAC | Baseline, 24 Weeks (Post Embolization Surgery)
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain index assesses participants' pain on a scale ranging from 0 (none) to 4 (extreme). The pain subscale consists of 5 items and total scores can range from 0-20, with larger scores indicating greater pain.
Incidence of treatment related adverse events | Up to 4 weeks (Post Embolization Surgery)
  Procedure-related and target knee osteoarthritis-related adverse events as assessed by treating physician

SECONDARY OUTCOMES:
Change in knee pain as assessed by VAS | Baseline, up to 52 weeks (Post Embolization Surgery)
  Visual Analog Scale (VAS) has a total score ranging from 0-10 with the higher score indicating greater pain
Change in knee pain | Baseline, up to 52 weeks (Post Embolization Surgery)
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain index assesses participants' pain on a scale ranging from 0 (none) to 4 (extreme). The pain subscale consists of 5 items and total scores can range from 0-20, with larger scores indicating greater pain.
Incidence of adverse events | Up to 52 weeks (Post Embolization Surgery)
  Procedure-related and target knee osteoarthritis-related adverse events as assessed by treating physician
WORMS Score for Synovitis | Baseline, up to 52 weeks (Post Embolization Surgery)
  Whole-Organ Magnetic Resonance Imaging Score (WORMS) has a score ranging from zero representing no knee problems and 332 representing knee problems
Kellgren-Lawrence Grade | Baseline, up to 52 weeks (Post Embolization Surgery)
  As assessed by X-Ray. Radiograph imaging graded on scale 1 (no arthritis) to 4 (severe arthritis)

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Ferreira De Souza, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No